CLINICAL TRIAL: NCT04779151
Title: An Open Label Phase II Basket Trial Exploring the Efficacy and Safety of the Combination of Niraparib and Dostarlimab in Patients With DNA Repair-deficient or Platinum-sensitive Solid Tumors
Brief Title: Basket Trial Exploring the Efficacy and Safety of the Combination of Niraparib and Dostarlimab
Acronym: NIRADO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Abandon of the partner, GSK
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-002766-14; 2020/3093 (Other: CSET number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Bladder Cancer; Gastric Adenocarcinoma; Gastro-oesophageal Adenocarcinoma; Head and Neck Cancer; Biliary Tract Cancer; Platinum-sensitive Urothelial Bladder Cancer; Clear Cell Renal Cell Carcinoma; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Biliary Tract Neoplasms; Carcinoma, Renal Cell | interventions — dostarlimab; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1.A - Urothelial Bladder Cancer (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Niraparib
- 1.B - Gastric or gastro-esophageal junction adenocarcinoma (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Niraparib
- 1.C - Head and Neck Cancer (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Niraparib
- 1.D - Biliary Tract Cancer and pancreatic ductal adenocarcinoma (PDAC) (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Niraparib
- 1.E - Others: any histology, excepted breast cancer, prostate cancer or serous ovarian cancer (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Niraparib
- Cohort 2 - Platinum-sensitive urothelial bladder cancer (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Niraparib
- Cohort 3 - Clear Cell Renal Cell Carcinoma (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Niraparib

INTERVENTIONS:
Drug: Dostarlimab — Substance: immunoglobulin G4 (IgG4) humanized monoclonal antibody (mAb) that binds with high affinity to PD-1 Manufacturer: Tesaro Inc. Dose: 500 mg every 21 days for the first 4 cycles, followed by 1,000 mg every 42 days cycle (ie, Q6W)
Drug: Niraparib — Substance: Inhibitor of poly-adenosine diphosphate [ADP] ribose polymerase (PARP) Manufacturer: Tesaro Inc. Dose: Flat-fixed dose (if <77kg or platelets <150,000 μL: 200mg; if >/=77kg and platelets >/= 150,000μL: 300mg)

SUMMARY:
Treatment will consist of a PARP inhibitor (niraparib) monotherapy priming period (cycle 0; 21 days); an anti-PD-1 antibody (Dostarlimab ; TSR-042) will then be added from C1D1 every 21 days in combination for the first 4 cycles, and then every 42 days. Disease will be assessed every 2 cycles (6 weeks) from C3D1 by CT-scan (or MRI or bone scan, if relevant). Patients still under treatment after 1 year may have tumor evaluation spaced out every 3 cycles

DETAILED DESCRIPTION:
This study will make it possible to evaluate the efficacy and safety of use of the combination of two products: niraparib and Dostarlimab (also called TSR-042). It will assess whether these two drugs can not only stop the growth of tumor cells but also activate immune cells to kill them.

Patients that tolerates these products well will also be monitored

The investigating doctor suggests that patient take part in this study because his disease may benefit from the treatments administered in this study. Only patients whose tumor is likely to respond to the drugs administered, based on preclinical results or clinical data, will be able to participate in this study. Patient are selected because his tumor seems to have the characteristics that allow him to be included in one of the following three cohorts:

Cohort 1: tumor has a particular mutation; this cohort will include 5 groups according to the type of cancer: bladder cancer (group 1A), cancer of the stomach or of the esophago-gastric junction (group 1B), head and neck cancer (group 1C), bile duct cancer (group 1D) or other cancers (group 1E) Cohort 2: tumor is bladder cancer and has shrunk under previous treatment with platinum salts Cohort 3: clear cell kidney cancer. These products have already been tested in combination and their combination has shown that it is possible without causing toxicity.

About 120 patients will participate in the study in several centers in France. All patients will receive the combination of these two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients must have histologically or cytologically confirmed progressive metastatic or recurrent solid tumor (as defined below for each tumor type). Diagnosis must be stated in a pathology report and confirmed by the physician investigator.
* Evidence of disease progression prior to trial entry.
* To be enrolled in this study, only the tumor types and settings described below are allowed:

4.1 - Cohorts 1 A-E: DNA repair deficiency, defined as bi-allelic loss-of-function alteration (mutation and/or deletion) in at least one of the following genes: ARID1A, ARID2, ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK2, FANCA, IDH1, IDH2, NBN, PALB2, PBRM1, RAD51C, RAD51D, FANCA, NBN, RAD51, RAD54L, SMARCA4.

4.1.1 - Cohort 1A: Urothelial Bladder Cancer

* Patients must have received at least one line of prior platinum - based systemic therapy. No more than 3 lines of previous systemic therapy for metastatic disease are allowed.

  * Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing platinum-based regimen is considered as first-line therapy.
  * Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the first-line therapy.
  * Patients must have platinum-sensitive disease defined as disease which reaches at least partial response after the last platinum chemotherapy line and the patient must have progressed at least 3 months after the last cycle of chemotherapy.
* Previous exposure to one line of anti-PD-1 or anti-PD-L1 is allowed, unless hyperprogression (Appendix 6) occurred on immunotherapy

4.1.2- Cohort 1B: Gastric or gastro-esophageal junction adenocarcinoma

* Metastatic or recurrent gastric or gastro-esophageal junction adenocarcinoma that has progressed following at least 1 and maximum 2 prior therapies, by imaging modalities.
* Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy is considered as first-line therapy.
* Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the first-line therapy.
* HER2-positive and -negative amplified patients are both eligible for entry into this study.
* Patients with HER2-positive gastric cancer must have received trastuzumab-containing regimen prior to study entry.
* Previous exposure to anti-PD-1 or anti-PD-L1 is not allowed

4.1.3- Cohort 1C: Head and Neck Cancer

* Histologically or cytologically confirmed carcinoma of the head and neck.
* Subjects are eligible regardless of HPV status
* Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy or chemo-radiotherapy regimen is considered as first-line therapy
* In case of previous platinum-based therapy, tumor progression or recurrence within 6 months of last dose of platinum-based therapy is not allowed.
* Previous exposure to one line of anti-PD-1 or anti-PD-L1 is allowed, unless hyperprogression (Appendix 6) occurred on immunotherapy
* Patients must have received at last one prior line of therapy in the advanced / metastatic setting
* No more than 2 lines of previous systemic therapy for metastatic disease are allowed.

4.1.4- Cohort 1D: Biliary Tract Cancer and pancreatic ductal adenocarcinoma (PDAC)

* Histologically or cytologically confirmed carcinoma of the biliary tract or PDAC that has progressed following at least 1 and maximum 2 prior therapies, by imaging modalities.
* Previous exposure to anti-PD-1 or anti-PD-L1 is not allowed

For PDAC only:

* Patients must have received at least 16 weeks of continuous first-line platinum-based chemotherapy without evidence of progression during that period
* Maximum of 1 prior line of therapy is allowed

4.1.5- Cohort 1E Others

* Any histology, excepted breast cancer, prostate cancer or serous ovarian cancer (Appendix 7).
* Previous exposure to one line of anti-PD-1 or anti-PD-L1 is allowed, unless hyperprogression (Appendix 6) occurred on immunotherapy 4.2 - Cohorts 2: Platinum-sensitive urothelial bladder cancer
* Patients must have received at least one line of prior platinum - based systemic therapy. No more than 3 lines of previous systemic therapy for metastatic disease are allowed.
* Platinum-sensitive disease is defined as disease which reached at least partial response after the last platinum chemotherapy line and progressed at least 3 months after the last cycle of chemotherapy
* Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing platinum-based regimen is considered as first-line therapy.
* Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the first-line therapy.
* Previous exposure to one line of anti-PD-1 or anti-PD-L1 is allowed, unless hyperprogression (Appendix 6) occurred on immunotherapy 4.3 - Cohort 3: Clear cell Renal Cell Carcinoma
* Patients must have received at least one line of previous therapy. No more than 4 previous lines of therapy are allowed.
* Patients must have received anti-PD-1 (or anti-PD-L1) in combination with an anti-CTLA-4 or an anti-angiogenic agent, and an antiangiogenic agent.
* Previous exposure to one line of anti-PD-1 or anti-PD-L1 is allowed unless hyperprogression (Appendix 6) occurred on immunotherapy For all cohorts: Representative archival formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (preferred) or 20 (ideally) freshly cut and unstained slides, with an associated pathology report, for ancillary studies and/or central testing. If less than 20 slides are available, inclusion must be discussed with the Coordinating Investigator. In all cases, recovery of the most recent tumor block or biopsy is encouraged. If no material is available (blocks or slides), a biopsy will be mandatory at baseline (before the start of the treatment).

For Cohorts 1A-E:

* For patients with DNA repair gene mutation already identified by local testing, mutational testing must have been done less than one year prior to inclusion in the trial (i.e. signing of informed consent). Tumor block should correspond to the one that has been used for the original testing. If no archival tissue available feasibility of a fresh tumor biopsy at baseline should be ensured and mutation confirmed on that tissue. Only tissue from core needle, punch or excisional biopsy sample collection will be accepted. Other methods such as fine-needle aspiration, brushing, bone tissue or lavage samples are not acceptable.
* For patients whose tissue will be evaluated by the Gustave Roussy DNA repair gene panel, original or more recent tumor blocks can be used.

  * At least one lesion, not previously irradiated, measurable according to RECIST v1.1) as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and suitable for repeated assessment.
  * Patients must have progressed following standard of care or not eligible to effective standard therapy
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration from registration date.
  * Estimated life expectancy of greater than 12 weeks.
  * Adequate hematologic and organ function, defined by the following laboratory results obtained within 3 days prior to the first study treatment (Cycle 0 Day 1):
  * Absolute neutrophil count (ANC) ≥ 1500 cells/μL (without granulocyte colony-stimulating factor support within 2 weeks before cycle 0 day 1).
  * Lymphocyte count ≥ 500/μL.
  * Platelet count ≥ 100.000/μL (without platelets transfusion within 2 weeks before Cycle 0 Day 1).
  * Hemoglobin ≥ 9g/dL (patients are not allowed to be transfused with RBC or receive erythropoietic treatment to meet this criterion).
  * Total bilirubin ≤ 1.5 ULN (subjects with documented/suspected Gilbert's disease or liver metastases may be enrolled with bilirubin ≤ 3 × ULN).
  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit (ULN) or ≤ 5 × ULN in case of liver involvement.
  * Albumin ≥ 28g/L.
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 40 mL/min (according to Cockroft and Gault formula).
  * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular weight heparin or warfarin) should be on stable dose.
  * Women of childbearing potential must have a negative serum β-HCG pregnancy test within 14 days prior to the administration of the first study treatment.Pregnancy testing must be repeated within 72 hours prior to the first dose and while on study.
  * Sexually active women of childbearing potential must agree to use a highly effective method of contraception supplemented by a barrier method, or to abstain from sexual activity during the study and for at least 180 days after the last study treatment administration.
  * Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.
  * Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
  * Sexually active males patients must agree to use condom during the study and for at least 180 days after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception for the same duration.
  * Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
  * Patient should be able and willing to comply with study visits and procedures as per protocol.
  * Patients must be affiliated to a social security system or beneficiary of an equivalent system.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product simultaneously and/or during the last 4 weeks (excepting observational or non-interventional clinical studies).
2. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug, or five half lives of the previous agent, whichever is the shorter.
3. Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks prior to Cycle 0 Day 1; or any radiation therapy within 1 week prior to Cycle 0 Day 1.
4. History of another primary malignancy within 5 years prior to Cycle 0 Day 1 except for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ without evidence of disease (eg, carcinoma in situ of the cervix, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).
5. Treatment with systemic corticosteroids or other immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor agents) within 2 weeks prior to Cycle 0 Day 1, or anticipated requirements for systemic immunosuppressive medications during the trial:

   o The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids for patients with orthostatic hypotension, low-dose supplemental corticosteroids for adrenocortical insufficiency and topical steroids for cutaneous diseases are allowed.
6. Acute toxicities from previous therapies that have not resolved to Grade ≤ 1, with the exception of alopecia.
7. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1.
8. Participant must not have received a platelet transfusion ≤ 4 weeks prior to Cycle 0 Day 1.
9. Participants must not have received colony stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior to Cycle 0 Day 1.
10. Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
11. Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
12. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
13. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the TSR-042 formulation, or to niraparib or its components.
14. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis.

    * Patients with autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible.
    * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible.
15. Active or prior documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis).
16. History of interstitial lung disease, idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia or evidence of active pneumonitis on screening chest CT scan.
17. History of allogeneic organ transplant or prior bone marrow transplantation of double umbilical cord blood transplantation.
18. Uncontrolled intercurrent illness including, but not limited to:

    * ongoing or active infection or severe infection requiring hospitalization or IV antibiotics within 2 weeks of starting treatment (with the exception of prophylactic antibiotics).
    * symptomatic congestive heart failure > NYHA II, superior vena cava syndrome, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, pericardial effusion, myocardial infarction within 90 days.
    * active peptic ulcer disease or gastritis.
    * active bleeding diatheses.
    * major seizure disorder
19. Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
20. Patients with known left ventricular ejection fraction (LVEF) < 40%; patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable cardiologic treatment.
21. Known positive test for HIV.
22. Patients with active hepatitis B (defined as positive HBsAg test at screening) or hepatitis C (HCV).Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen anti-HBc) are eligible.
23. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
24. Active tuberculosis.
25. Administration of attenuated or live vaccine within 4 weeks prior to Cycle 0 Day 1 or anticipation that such a live attenuated vaccine will be required during the study.
26. Major surgical procedure within 20 days prior ty Cycle 0 Day 1 or anticipation of need for a major surgical procedure during the course of the study.
27. Uncontrolled tumor-related pain: patients requiring pain medication must be on a stable regimen at study entry and symptomatic lesions amenable to palliative radiotherapy should be treated prior to enrolment.
28. Uncontrolled effusion (pleural, pericardial or ascites) requiring recurrent drainage procedures (once a month or more frequently); patients with indwelling catheters (e.g. PleurX) are allowed.
29. Uncontrolled hypercalcemia (>1.5mmol/L ionized calcium or Ca > 12mg/dL or corrected serum calcium >ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.

    * Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history or clinically significant hypercalcemia are eligible.
    * Patients who are receiving denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate instead while on study.
30. History of leptomeningeal disease

    * Symptomatic CNS metastasis or uncontrolled CNS metastasis, requiring increasing doses of steroids or stable dose of steroids > 10mg prednisone qd.
    * Spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to Cycle 0 Day 1.
31. Previous treatment with PARP inhibitors.
32. Treatment with systemic immunostimulatory agents (e.g. INF-a and IL-2) within 4 weeks prior to Cycle 0 Day 1.
33. Patients with rare hereditary problems of galactose intolerance, the lapp lactase deficiency or glucose galactose malabsorption
34. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study result.
35. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | at 15 weeks
  according to Response Evaluation Criteria In Solid Tumors v1.1 (RECIST v1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

IPD SHARING:
Plan to Share IPD: No